CLINICAL TRIAL: NCT05680350
Title: Plasma Levels of Micro RNA 203 and 210 Might Spare the Exploratory Laparoscopy in Case of un Explained Infertility With Suspected Endometriosis
Brief Title: Relation Between MicroRNA 203 and 210 and Sparing the Laparoscopic Examination in Cases of Unexplained Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Amr Sharaf Eldein, Assistant professor of gynecology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RC 2.6.2022
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Infertility Unexplained; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Study group Patients with unexplained infertility had estimated their Plasma Expression level for Gene"Micro RNA "203 & 210" by qRT-PCR followed by laparoscopic exploration
  Interventions: Procedure: Laparoscopic Exploration; Diagnostic Test: Estimation of Plasma Expression level of MICRO RNA 203 & 210
- Control Group (Active Comparator): Control group Patients with unexplained infertility underwent laparoscopy only
  Interventions: Procedure: Laparoscopic Exploration

INTERVENTIONS:
Procedure: Laparoscopic Exploration — Laparoscopic Exploration to diagnose & grade endometriosis
Diagnostic Test: Estimation of Plasma Expression level of MICRO RNA 203 & 210 — estimation of Plasma Expression level for Gene"Micro RNA "203 & 210" by qRT-PCR
  Arms: Study group

SUMMARY:
The study targets to evaluate the role of estimation of plasma expression levels of gene of microRNAs 203 and 210 in helping to diagnose and grade endometriosis. The study included women with unexplained infertility and clinical picture suggestive of presence of endometriosis were divided randomly into two groups: Control and study groups. All patients underwent exploratory laparotomy for diagnosis and grading of endometriosis if present. Patients of study group gave blood samples for estimation of plasma expression levels of microRNA 203 and 210 using qRT-PCR procedure.

ELIGIBILITY:
Inclusion Criteria:

* 30-45 years old
* Unexplained infertility

Exclusion Criteria:

* Presence of other causes of infertility,
* age out of the predetermined range,
* the presence of immune disorders,
* maintenance on immunosuppressive drugs

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-11-07 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
grading of endometriosis | 8 months
  The diagnostic performance of estimated plasma levels of microRNA for diagnosis and grading endometriosis

CONTACTS AND LOCATIONS:
Locations (1):
- Banha University, Banhā, El- Qalyobia, Egypt